CLINICAL TRIAL: NCT02409394
Title: Effect of a High-fat Meal on the Pharmacokinetics of Hetrombopag and Mass Balance Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TPOP1c
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hetrombopag 7.5mg fasted to fed (Experimental): Hetrombopag tablet, fasting conditions on day 1; 9 days wash-out; Than subjects will be crossover to have hetrombopag tablet with high fat, high calorie breakfast on day 11.
  Interventions: Drug: Hetrombopag Olamine
- hetrombopag 7.5mg fed to fasted (Experimental): Hetrombopag tablet with high fat, high calorie breakfast on day 1; 9 days wash-out; Than subjects will be crossover to have hetrombopag tablet, under fasting condition on day 11.
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine

SUMMARY:
This open-label, randomized, two-period, two-treatment (single doses of 7.5 mg hetrombopag fasted or fed), crossover study was conducted to evaluate the effect of a high-fat meal on the pharmacokinetics of hetrombopag and mass balance study in 12 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Weight≥50 kg，19≤BMI≤28 kg/m2.
* Platelet count is within normal range

Exclusion Criteria:

* History of clinically significant illness.
* History of alcohol or drug abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of hetrombopag | 0h-120h
  Cmax (a measure of the body's exposure to hetrombopag) will be compared under fating state and fasted state
The area under the plasma concentration-time curve (AUC) of hetrombopag | 0h-120h
  AUC (a measure of the body's exposure to hetrombopag) will be compared under fating state and fasted state
The accumulative excretion rate of hetrombopag and its metabolites in urine and feces | 0h-120h

SECONDARY OUTCOMES:
The change of platelet count | On day 2, 4, 6, 8,12, 14 and 16
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 16

CONTACTS AND LOCATIONS:
Locations (1):
- West Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Wang Z, Chen X, Li A, Chen L, Wang Y, Zheng L. Effect of Food on the Pharmacokinetic and Pharmacodynamic Profiles of Hetrombopag in Healthy Volunteers. Clin Ther. 2020 Dec;42(12):2280-2288. doi: 10.1016/j.clinthera.2020.10.002. Epub 2020 Oct 24. PMID 33109386